CLINICAL TRIAL: NCT01317290
Title: Accumulation of n-3 Long-chain (LC)-PUFA by Supplementation of ALA-rich Oil in Humans Depending on Age, Gender and Physiological Stage.
Brief Title: Supplementation of Alpha-linolenic Acid (ALA)-Rich Oil in Humans
Acronym: ALA_KK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil., University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H50-11-KK
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Overweight; Hypercholesterolemia
Keywords: Conversion of ALA
MeSH Terms: conditions — Overweight; Hypercholesterolemia | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- linseed oil; young (Experimental): ALA rich linseed oil to younger subjects (18-35 years)
  Interventions: Dietary Supplement: linseed oil
- linseed oil; older (Experimental): ALA rich linseed oil to older, normalweight subjects (BMI <25, age 49-69 years)
  Interventions: Dietary Supplement: linseed oil
- linseed oil older, overweight (Experimental): ALA-rich linseed oil to older, normalweight subjects (BMI >25, age 49-69 years)
  Interventions: Dietary Supplement: linseed oil
- olive oil (Experimental): n3-PUFA free control oil to normalweight subjects (BMI <25)
  Interventions: Dietary Supplement: n-3 PUFA free olive oil

INTERVENTIONS:
Dietary Supplement: n-3 PUFA free olive oil — negative control
  Arms: olive oil
Dietary Supplement: linseed oil
  Arms: linseed oil older, overweight; linseed oil; older; linseed oil; young

SUMMARY:
The objective of this study is to investigate the accumulation of n-3 LC-PUFA (EPA, DPA and DHA) in human lipids by oral supplementation of ALA-rich linseed oil. In addition, the accumulation of n-3 LC-PUFA is compared between subpopulations of different age, gender and physiological conditions (overweight, increased serum total cholesterol).

DETAILED DESCRIPTION:
N-3 PUFA are important for human health and nutrition. Unfortunately, the land-based n-3 ALA is a limited precursor for the formation of n-3 LC-PUFA. The conversion of ALA depends on the rate-limiting ∆6-desaturation.

The first objective of this study is to investigate differences of the accumulation of n-3 LC-PUFA (EPA, DPA and DHA) in human lipids during supplementation of ALA-rich linseed oil dependent on age, gender and physiological conditions (overweight, increased serum total cholesterol). One study group will receive fish oil with mainly EPA as positive control.

The second objective is to compare the n-3 LC-PUFA enrichment during the linseed oil supplementation (study LSEP H50-KK) with the n-3 LC-PUFA enrichment during the further Echium oil supplementation (study LSEP H42-KK). The second study will be the control for the first study.

Therefore, it is planned to recruit the same subjects for the linseed oil supplementation.

Eighty volunteers will be recruited and allocated into four study groups depending on age and BMI. Three groups (each n=20) will receive daily ca. 15 g linseed oil (mean age: 25 and 55 years; mean BMI < 25; and mean age 55 and BMI > 25). One group (n=20) will receive n-3PUFA free olive oil (mean age 25 and 55, BMI < 25). The double-blind, randomized, parallel-designed study will start with a two-weeks run-in period, followed by an eight-weeks supplementation period. After the run-in period, one week and eight weeks of oil supplementation blood will be drawn and 24-h urine will be sampled.

Altogether, the fatty acid distribution after Echium oil and linseed oil supplementation from similar subjects can be statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* cholesterol lowering drugs
* chronic diseases
* pregnancy, lactation
* intake of nutritional supplements

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
n-3 LC-PUFA in human lipids (EPA) | 0,7,56 days
  EPA (% of total identified fatty acid methyl esters)

SECONDARY OUTCOMES:
eicosanoid concentration in plasma | 0 and 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Kuhnt, Dr. rer. nat, Principal Investigator — University of Jena, Insitute of Nutrition
Locations (1):
- Friedrich Schiller University of Jena, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Kuhnt K, Weiss S, Kiehntopf M, Jahreis G. Consumption of echium oil increases EPA and DPA in blood fractions more efficiently compared to linseed oil in humans. Lipids Health Dis. 2016 Feb 18;15:32. doi: 10.1186/s12944-016-0199-2. PMID 26892399
- [Derived] Grindel A, Staps F, Kuhnt K. Cheek cell fatty acids reflect n-3 PUFA in blood fractions during linseed oil supplementation: a controlled human intervention study. Lipids Health Dis. 2013 Nov 14;12:173. doi: 10.1186/1476-511X-12-173. PMID 24229084